CLINICAL TRIAL: NCT06822283
Title: Investigation of the Plasticity of Deep Brain Structures in Mild Cognitive Impairment and Healthy Aging (PlasMA)
Brief Title: Plasticity of Deep Brain Structures in Mild Cognitive Impairment and Healthy Aging
Acronym: PlasMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedhelm Hummel (Other)
Collaborators: Clinique Romande de Readaptation (Network); HUG University hospital (Unknown); SNF Swiss National Foundation (Unknown); The Novartis Foundation (Other); Fondation Bertarelli (Unknown); Wyss Center for Bio and Neuroengineering (Other)
Responsible Party: Sponsor-Investigator, Friedhelm Hummel, Prof. Dr. med., Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-00127
Record Dates: First submitted 2025-01-13; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Traumatic Brain Injury
Keywords: non-invasive brain stimulation; deep brain stimulation; subcortical; memory; neuro-imaging; transcranial temporal interference stimulation; motor learning
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo stimulation (Placebo Comparator): Sham stimulation : ramp-up [5 s] immediately followed by ramp-down [5 s] of high-frequency currents (see Vassiliadis et al., 2023, Nat Hum Behav for more details)
  Interventions: Other: transcranial electric stimulation
- Active stimulation (Experimental): Patterned stimulation (intermittent theta-burst) generating temporal interference in the striatum; see Wessel et al., 2023, Nat Neurosci. for details
  Interventions: Other: transcranial electric stimulation

INTERVENTIONS:
Other: transcranial electric stimulation — tTIS is an innovative non-invasive brain stimulation approach, in which two or more independent stimulation channels deliver high-frequency currents in the kHz range (oscillating at f1 and f1 + Δf). These high-frequency currents are assumed to be too high to effectively modulate neuronal activity. Still, by applying a small shift in frequency, they result in a modulated electric field with the envelope oscillating at the low-frequency Δf (target frequency) where the two currents overlap. The peak of the modulated envelope amplitude can be steered towards specific areas located deep in the brain, by tuning the positions of the electrodes and the current ratio across stimulation channels. Here, we applied tTIS via surface electrodes applying a low-intensity (2mA baseline to peak), sub-threshold protocol following the safety guidelines for low-intensity transcranial electric stimulation in humans.

SUMMARY:
Acute and chronic cognitive impairment (TBI and MCI) is one of the most common problems in the growing and aging society of the 21st century. At an individual level, not all brain structures are affected with the same rate. There are subcortical structures less involved (e.g., the cerebellum), and other more involved (e.g., the hippocampus) in the cognitive decline with age or following a traumatism. To pave the way for personalized precision medicine in the field of cognitive preservation and recovery, there is a need for testing the impact of individually tailored innovative non-invasive neuro-technologies. In this project, we aim at testing the benefit of non-invasively stimulating subcortical structures to boost resilience in supporting motor and non-motor memory.

ELIGIBILITY:
Inclusion Criteria:

TBI patients:

* Age ≥ 18 years
* Clinical diagnosis of TBI
* No history of other severe neurological or psychiatric disorders

Exclusion Criteria:

* Unable to consent

  * Severe neuropsychiatric (e.g., major depression, severe dementia) or unstable systemic diseases (e.g., severe progressive and unstable cancer, life threatening infectious diseases)
  * Severe sensory or cognitive impairment or musculoskeletal dysfunctions prohibiting to understand instructions or to perform the experimental tasks
  * Inability to follow or non-compliance with the procedures of the study
  * Contraindications for NIBS or MRI (1):

    * Electronic or ferromagnetic medical implants/device, non-MRI compatible metal implant
    * History of seizures
    * Medication that significantly interacts with NIBS being benzodiazepines, tricyclic antidepressants and antipsychotics
  * Regular use of narcotic drugs
  * Pregnancy
  * Request of not being informed in case of incidental findings
  * Concomitant participation in another trial involving probing of neuronal plasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Motor learning performance | From baseline to 24 hours after training
  The primary outcome of the study is the amount of motor learning in a sequential finger-tapping task evaluated during and following training

SECONDARY OUTCOMES:
Brain connectivity | Baseline measure (before the intervention)
  Diffusion-weighted and resting-state MRI is performed at baseline and allows to evaluate inter-individual anatomical factors associated to the primary outcome

OTHER OUTCOMES:
Demographic factors form | Baseline measure (before the intervention)
  These factors including age, sex, handedness, education level and profession, time of diagnosis, physical activity, independency and quality of life, medication, cognitive status will are used to evaluate responsiveness to the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - EPFL Valais, Clinique Romande de readaptation, Sion, Valais
  - EPFL, Campus Biotech, Geneva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wessel MJ, Beanato E, Popa T, Windel F, Vassiliadis P, Menoud P, Beliaeva V, Violante IR, Abderrahmane H, Dzialecka P, Park CH, Maceira-Elvira P, Morishita T, Cassara AM, Steiner M, Grossman N, Neufeld E, Hummel FC. Noninvasive theta-burst stimulation of the human striatum enhances striatal activity and motor skill learning. Nat Neurosci. 2023 Nov;26(11):2005-2016. doi: 10.1038/s41593-023-01457-7. Epub 2023 Oct 19. PMID 37857774
- [Background] Vassiliadis P, Beanato E, Popa T, Windel F, Morishita T, Neufeld E, Duque J, Derosiere G, Wessel MJ, Hummel FC. Non-invasive stimulation of the human striatum disrupts reinforcement learning of motor skills. Nat Hum Behav. 2024 Aug;8(8):1581-1598. doi: 10.1038/s41562-024-01901-z. Epub 2024 May 29. PMID 38811696
- [Result] Vassiliadis P, Stiennon E, Windel F, Wessel MJ, Beanato E, Hummel FC. Safety, tolerability and blinding efficiency of non-invasive deep transcranial temporal interference stimulation: first experience from more than 250 sessions. J Neural Eng. 2024 Mar 11;21(2). doi: 10.1088/1741-2552/ad2d32. PMID 38408385